CLINICAL TRIAL: NCT07341360
Title: Pseudovav - A Cancer Vaccine Targeting Mutated GNAS Combined With Immune Checkpoint Inhibition for Patienes With Pseudomyxoma Peritonei
Brief Title: Pseudovax - A Cancer Vaccine for Patients With Pseudomyxoma Peritonei
Acronym: Pseudovax
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Geir Olav Hjortland, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-517047-30-01; 2024-517047-30-01 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pseudomyxoma Peritonei
Keywords: Pseudovax; PMP; Peptide vaccine; GNAS mutation; pseudomyxoma peritonei
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — molgramostim; tislelizumab

STUDY DESIGN:
Intervention Model Description: Study Design: A phase 1, first-in-human open label, single-arm trial, combining the novel peptide vaccine Pseudovax against mutated GNAS (Gsα) with adjuvant granulocyte macrophage - colony stimulating factor (GM-CSF) and subsequent treatment with the immune checkpoint inhibitor tislelizumab (anti-PD-1) in adult subjects with recurrent or non-resectable GNAS-mutated pseudomyxoma peritonei (PMP).
  Study treatment: Participants will be administered the Pseudovax peptide vaccine + adjuvant, granulocyte-macrophage colony-stimulating factor (GM-CSF). From study week 13, the programmed cell death 1 (PD-1) inhibitor tislelizumab will be administered in addition, for a maximum of 21 months, until confirmed progression, unacceptable toxicity, withdrawal of consent, or Investigator decision, whichever happens first.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pseudovax peptide, adjuvant and PD-1 inhibitor (Experimental): Participants will be administered the Pseudovax peptide vaccine + adjuvant, granulocyte-macrophage colony-stimulating factor (GM-CSF). From study week 13, the programmed cell death 1 (PD-1) inhibitor tislelizumab will be administered in addition, for a maximum of 21 months, until confirmed progression, unacceptable toxicity, withdrawal of consent, or Investigator decision, whichever happens first.
  Interventions: Other: Pseudovax; Biological: Molgramostim; Biological: Tislelizumab

INTERVENTIONS:
Other: Pseudovax — Pseudovax peptide dissolved in 0.5 mL water for injection to 1 mg/mL (+/- 0.1 mg/mL)
Biological: Molgramostim — Molgramostim, 100 μg recombinant human GM-CSF, powder, to be reconstituted in 0.33 mL water for injection
Biological: Tislelizumab — 100 mg of humanized IgG4 mAb in 10 mL of isotonic solution

SUMMARY:
Participants will receive vaccination with Pseudovax/GM-CSF in combination with PD-1 inhibitor tislelizumab over a period of up to two years. The vaccine is expected to reactivate measurable immune response, and tislelizumab to restore anticancer immunity in patients with GNAS mutated pseudomyxoma peritonei.

DETAILED DESCRIPTION:
Pseudomyxoma peritonei (PMP) is a rare, slow-growing abdominal cancer that commonly originates in ruptured appendiceal mucinous neoplasms, which seed tumor cells and mucin into the peritoneal cavity. The disease is characterized by slow, progressive growth and accumulation of mucinous tumor tissue in the peritoneal cavity, ultimately leading to abdominal compression and death. Standard-of-care treatment (SOC) involves extensive cytoreductive surgery (CRS) followed by hyperthermic intraperitoneal chemotherapy (HIPEC), and is curative in approximately 50% of the patients, but for patients who cannot be cured by SOC, no efficacious treatment options exist. In the setting of non-resectable and recurrent disease, PMP is a debilitating and ultimately fatal condition, leaving patients to experience progressively poor quality of life caused by an increasing intraperitoneal tumor burden. In research carried out by the study team, mutated GNAS as a potential tumor neo-antigen was investigated by analyzing tumor and peripheral blood samples collected from PMP patients at the time of surgery.

The results (detailed in the Pseudovax IB) indicated that the patients had a strong immune response against mutated GNAS. However, the presence of a high tumor burden at the time of surgery implies that the immune response had been insufficient to control tumor growth. Further analyses revealed that this could be explained by inhibition of anti-tumor T cells by up-regulation of immune checkpoint molecules.

These results provide the rationale for vaccination targeting mutated GNAS to increase the number of tumor cell targeting T cells. Furthermore, the observed up-regulation of programmed death-1 (PD-1) on intratumoral T cells provides rationale for combining the vaccination with a PD-1 inhibitor. Importantly, very few patients with PMP have had the opportunity to test treatment with immune checkpoint inhibitors. The main reason is that PMP molecularly is a microsatellite stable disease with very low tumor mutational burden, and patients are therefore not likely to respond to immune-check point inhibition (ICI) monotherapy. The planned combination with the Pseudovax peptide vaccine may represent a unique opportunity to derive benefit from ICI treatment for this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is ≥ 18 years of age on the day of signing the informed consent form, able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
2. Confirmed diagnosis of recurrent or non-resectable PMP with no other available treatment options that are expected to be efficacious.
3. The subject's tumor must carry a mutation in the GNAS oncogene*
4. Subjects must have peritoneal tumor distribution at screening that, in the opinion of the Investigator, is suitable for repeat biopsies: Up to 3 biopsies of target tissue are planned for subjects that complete the study.
5. Adequate organ, bone marrow, liver, and renal function at screening, including:

   1. Absolute neutrophil count: ≥ 1,5 x109/L
   2. Platelets: ≥ 100 x109/L
   3. Hemoglobin: ≥ 9 x109/L
   4. Creatinine ≤ 1,5 upper limit normal (ULN) OR measured/calculated GFR ≥60 mL/min
   5. Albumin ≥ 30 g/L
   6. Total bilirubin ≤ 1,5 ULN
   7. ASAT and ALAT ≤ 3 ULN
   8. International Normalized Ratio (INR) ≤ 1,5 ULN and Activated Partial Thromboplastin Time (aPTT) ≤ 1,5 ULN unless subject is receiving anticoagulant therapy.
6. ECOG performance status of 0 or 1.
7. Life expectancy of >6 months, at the time of signing the informed consent.
8. Women of childbearing potential must have a negative serum pregnancy test within 48 hours of the first study intervention, and must not be breast-feeding. 8ai. Female participant:

   i. Unless documented not to have childbearing potential: Subject is willing to use contraceptive measures for the duration of the study, and ≥ 6 months after the last dose of IMP, as prescribed by the protocol (according to the applicable guidance: CTFG, 2020). The Investigator should counsel women of childbearing potential of the importance of pregnancy prevention.

8aii. Women of childbearing potential must have a negative serum pregnancy test within 48 hours of the first study intervention.

8b. Male subject: Sexually active males must be willing to use a condom during sex for the duration of the study and for ≥ 6 months after the last dose of IMP. Males must also be willing to abstain from donating sperm during the same period.

Exclusion Criteria:

1. Patient has Eastern Cooperative Oncology Group performance status 2 or worse.
2. Blood transfusion or growth factor support ≤ 14 days before sample collection at screening.
3. Active malignancy the past 3 years except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
4. Enrollment in another interventional trial that, in the opinion of the Investigator, could influence the outcome of this study.
5. Subject has within the last 30 days received any other interventional therapy that, in the opinion of the Investigator, could influence the outcome of this study.
6. Pregnancy or lactating female.
7. Known active hepatitis B or C, or is known to be HIV-positive.
8. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of IMP.

   Note: Subjects who are currently or have previously been on any of the following steroid regimens are not excluded: Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent); Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption; Short course (≤ 7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen).
9. Active autoimmune diseases or history of autoimmune diseases that may relapse. Note: Subjects with the following diseases are not excluded and may proceed to further screening, controlled Type I diabetes, hypothyroidism (provided it is managed with hormone replacement therapy only), controlled celiac disease skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia), any other disease that is not expected to recur in the absence of external triggering factors.
10. Diagnosis of immunodeficiency.
11. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
12. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.
13. Severe infections within 4 weeks before first dose of IMP, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
14. Therapeutic oral or intravenous antibiotics within 2 weeks before first dose of IMP.
15. Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of IMP.
16. Prior allogeneic stem cell transplantation or organ transplantation
17. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of IMP.
18. Pulmonary embolism ≤ 28 days before first dose of IMP.
19. History of acute myocardial infarction ≤ 6 months before first dose of IMP.
20. History of heart failure meeting New York Heart Association (NYHA) Classification III or IV (Appendix 6) ≤ 6 months before first dose of IMP.
21. Subject has had any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before first dose of IMP.
22. Severe hypersensitivity (≥grade 3) to chemotherapy, any other biologic drug or the contents or preservatives of any of the study drugs.
23. History of cerebrovascular accident ≤ 6 months before first dose of IMP.
24. Subject has underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct.
25. Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of sequential treatment with Pseudovax/GM-CSF and tislelizumab | From start treatment to 6 months after last dose of study drug.
  Incidence of Investigative Medicinal Product-related adverse events. All ≥ Grade 3 adverse events and all grades vaccine-related adverse events will be reported and graded using CTCAE v 5.0.
Immune responses following sequential treatment with Pseudovax/GM-CSF and tislelizumab | From enrollment to end of treatment (2 years).
  Count of circulating vaccine-specific T cells

SECONDARY OUTCOMES:
Progression-free survival, measured as the number of months from date of first treatment until disease progression or death from any cause | From start treatment to disease progression, death or last follow-up 6 months after last dose of study drug (whichever comes first).
  Assessment of preliminary efficacy of study treatment with Pseudovax/GM-CSF and Tislelizumab, measured as the number of months from date of first treatment until disease progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital HF, Radium, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
By now there is no plan on sharing IPD as the patient group is very small (ten patients plan) with a rare disease. As a result we can not make this data widely available without violating GDPR guidance. For researchers interested in the data, a request can be send to the study team.